CLINICAL TRIAL: NCT05855863
Title: Clinical Study of Ginkgo Biloba Ketone Ester Tablets in Diabetes Related Dementia
Brief Title: Clinical Study of GKT in Diabetes Related Dementia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Guoxiang Fu, Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GKT
Record Dates: First submitted 2023-04-10; First posted 2023-05-12 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ginkgo Ketone Ester Tablets Treatment Group (Experimental): Ginkgo Ketone Ester Tablets (Styron), taken orally, 3 times a day, 0.5g each time, combined with conventional hypoglycemic therapy continuously administered for 6 months
  Interventions: Drug: Ginkgo Ketone Ester Tablets
- control group (Placebo Comparator): placebo combined with conventional hypoglycemic therapy for 6 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ginkgo Ketone Ester Tablets — Ginkgo Ketone Ester Tablets taken orally, 3 times a day, 0.5g each time, combined with conventional hypoglycemic treatment for six months
  Other Names: Test group
  Arms: Ginkgo Ketone Ester Tablets Treatment Group
Drug: placebo — placebo, taken orally, 3 times a day, 0.5g each time, combined with conventional hypoglycemic treatment for six months
  Other Names: Control group
  Arms: control group

SUMMARY:
Recently a new clinical dementia subgroup based on brain imaging, called "diabetes related dementia (DrD)". DrD, unlike Alzheimer's disease and vascular dementia, is considered a "controllable" or "modifiable" form of dementia. However, there is currently a lack of corresponding treatment measures. Ginkgo biloba ketone ester tablets are extracts of Ginkgo biloba leaves. Previous studies have shown that they can increase cerebral blood flow, reduce cerebrovascular resistance, improve cerebral circulation, and are beneficial for the treatment of cognitive impairment. This project intends to explore the role of ginkgo ketoester tablets in diabetes related dementia through a multicenter randomized double-blind controlled clinical study.

DETAILED DESCRIPTION:
This study was divided into two treatment groups: the experimental group and the control group. 370 type 2 diabetes patients with mild cognitive impairmentpatients were randomly selected and assigned to the experimental group of 185 patients and the control group of 185 patients in a 1:1 equal amount. Experimental group: Ginkgo biloba ketone ester tablets combined with conventional hypoglycemic treatment group, the usage is Ginkgo biloba ketone ester tablets (Styron), taken orally, 3 times a day, 0.5g each time, and continuously administered for 6 months. Control group: conventional hypoglycemic treatment group. The Montreal Cognitive Assessment Basic (MoCA-B) was used for the detection of cognitive dysfunction. Neuropsychological testing of cognitive function was conducted using Alzheimer's Disease Assessment Scale - Cognitive Scale (ADAS-cog), Auditory Word Learning Test (AVLT-H);Assessment of Daily Living Ability - Functional Activity Questionnaire (FAQ);Shape Connection Test A and B and Symbolic Digital Form Test (SDMT).Collect patients' blood, and detect C-reactive protein, interleukin-6, oxidative stress, ApoE4 genotype, phosphorylated tau protein, irisin, β- Amyloid protein before and after the experiment.Detect changes in ankle brachial pulse wave conduction velocity (baPWV)/and ankle brachial blood pressure index (ABI) of patients before and after the experiment.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes with mild cognitive impairment patients aged 65 years or above;
2. Able to cooperate in completing cognitive function testing;
3. Patients who can swallow pills
4. No previous history of stroke，cerebral thrombosis, etc

Exclusion Criteria:

1. Type 1 diabetes;
2. Acute cerebral infarction and myocardial infarction within 3 months;
3. Severe liver and kidney dysfunction;
4. Late stage malignant tumors;
5. Thyroid dysfunction；
6. Brain injury and cerebral hemorrhage within 3 months；
7. Folic acid and/or vitamin B12 deficiency
8. Patients who are currently using thrombin inhibitors, defibrillators (with unclear efficacy in ischemic stroke and increased risk of bleeding), antiplatelet drugs, blood activating and stasis resolving agents, and other ginkgo biloba leaf preparations (as they may affect the evaluation of the therapeutic effect of ginkgo biloba ester tablets in this trial), as well as other trial medications.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function testing | six months
  Alzheimer's Disease Assessment Scale-Cognitive section (0-70), the higher the score, the more severe the cognitive impairment

SECONDARY OUTCOMES:
Memory function assessment | six months
  Auditory Word Learning Test (AVLT-H),the lower the score, the more severe the cognitive impairment
Assessment of daily living ability | six months
  Functional Activity Questionnaire (FAQ)S,the higher the score, the more severe the cognitive impairment
Perform functional evaluation | six months
  Shape Connection Test A and B (STT-A&B)，the higher the score, the more severe the cognitive impairment
Attention assessment | six months
  Symbolic Digital Form Test (SDMT)，the lower the score, the more severe the cognitive impairment

OTHER OUTCOMES:
Concentration of C-reactive protein | six months
  Human CRP(C-Reactive Protein) ELISA Kit for detecting C-reactive protein concentration (mg/L )in serum
Rate of arteriosclerosis in the large and middle arterial systems | six months
  ankle brachial pulse wave conduction velocity (m/s )detected by Arteriosclerosis tester
Rate of arterial blockage in limbs | six months
  ankle brachial blood pressure index (ABI) measures ankle blood pressure and upper arm brachial artery blood pressure through ankle brachial index instrument
Concentration of interleukin-6 | six months
  interleukin-6(IL-6) in serum detected by interleukin-6 ELISA Kit
Concentration of phosphorylation (p) - tau217 | six months
  Plasma phosphorylation (p) - tau217detected by P-Tau217 detection kit
Concentration of Amyloid protein Aβ 42/40 | six months
  Plasma Amyloid protein Aβ 42/40 detected by Aβ 42/40 detection kit
Participants with ApoE4 genotype | six months
  ApoE4 genotype detected by ApoE4 genotype kit
Concentration of antioxidant enzyme activity | six months
  Detection of glutathione peroxidase in serum
Concentration of oxidative stress | six months
  Free radical detection in serum
Concentration of irisin | six months
  Plasma irisin concentration detected by irisin ELISA kit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fukazawa R, Hanyu H, Sato T, Shimizu S, Koyama S, Kanetaka H, Sakurai H, Iwamoto T. Subgroups of Alzheimer's disease associated with diabetes mellitus based on brain imaging. Dement Geriatr Cogn Disord. 2013;35(5-6):280-90. doi: 10.1159/000348407. Epub 2013 Apr 13. PMID 23594859
- [Result] Hanyu H, Hirose D, Fukasawa R, Hatanaka H, Namioka N, Sakurai H. Guidelines for the Clinical Diagnosis of Diabetes Mellitus-Related Dementia. J Am Geriatr Soc. 2015 Aug;63(8):1721-3. doi: 10.1111/jgs.13581. No abstract available. PMID 26289708
- [Result] Verdile G, Fuller SJ, Martins RN. The role of type 2 diabetes in neurodegeneration. Neurobiol Dis. 2015 Dec;84:22-38. doi: 10.1016/j.nbd.2015.04.008. Epub 2015 Apr 26. PMID 25926349
- [Result] Fukasawa R, Hanyu H, Namioka N, Hatanaka H, Sato T, Sakurai H. Elevated inflammatory markers in diabetes-related dementia. Geriatr Gerontol Int. 2014 Jan;14(1):229-31. doi: 10.1111/ggi.12140. No abstract available. PMID 24405824
- [Result] Hatanaka H, Hanyu H, Fukasawa R, Sato T, Shimizu S, Sakurai H. Peripheral oxidative stress markers in diabetes-related dementia. Geriatr Gerontol Int. 2016 Dec;16(12):1312-1318. doi: 10.1111/ggi.12645. Epub 2015 Nov 4. PMID 26531676
- [Result] Hirose D, Hanyu H, Fukasawa R, Hatanaka H, Namioka N, Sakurai H. Frailty in diabetes-related dementia. Geriatr Gerontol Int. 2016 May;16(5):653-5. doi: 10.1111/ggi.12566. No abstract available. PMID 27109174